CLINICAL TRIAL: NCT05130723
Title: Pharmacokinetics of Fluconazole Given Orally or Intravenously as Prophylaxis or Therapy to Children and Adolescents With Invasive Fungal Infections
Brief Title: Pharmacokinetics of Fluconazole in Children (2-18 Years)
Acronym: FOCUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF-21.05; 2021-006868-24 (EudraCT Number)
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Invasive Fungal Infections
Keywords: Pharmacokinetics; Antifungal drugs; Pediatrics
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be obtained an processed to obtain plasma. Fluconazole plasma levels will be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Pediatric patients aged 2-18 years administered with fluconazole for the treatment or prophylaxis of invasive fungal infections.

SUMMARY:
30 pediatric patients aged 2-18 years receiving fluconazole as part of standard care for the treatment or prophylaxis of an invasive fungal infection will be included in the study. Between day 2 and 10, 6 samples will be collected on two days. In the case a patient switches from oral to intravenous therapy, an additional PK-day consisting of 3 samples will be scheduled. Fluconazole plasma concentrations will be determined. A pharmacokinetic model will be fitted to the data from all individuals simultaneously. Data will be analysed using non-linear mixed effects modelling (NONMEM). Monte Carlo simulations will guide the establishment of an improved fluconazole dosing regimen for pediatric and adolescent patients.

DETAILED DESCRIPTION:
Fluconazole has been available since 1990, however a limited number of studies addressed the pharmacokinetics (PK) of fluconazole in children and adolescent patients. Solid PK data are lacking, despite there being expected variation due to physiological differences with adults likely resulting in significant clinical impact. Especially in the paediatric population where fluconazole is extensively used, including in patients who have moderate to severe renal function disturbances, this information is needed. Therefore, it seems prudent to conduct a study in a cohort of paediatric patients who receive fluconazole as prophylaxis or treatment. The primary objective of the study is to establish an improved fluconazole dosing regimen for paediatric and adolescent patients aged 2-18 years.

A total of pediatric 30 patients will be included in this observational PK-study. Patients will receive standard fluconazole therapy according to (local) protocol. Blood samples will be collected from already placed arterial or central venous catheter.

Between day 2 and 10, six blood samples will be collected for the purpose of PK analysis. Samples will be collected on two different days. On the first PK-day, 3 samples will be collected on t = 0, 1, and 5 hours after fluconazole administration and on the second PK-day, 3 samples will be collected on t = 0.5, 3, and 7 hours after fluconazole administration.

If the patient is expected to switch from iv to oral therapy or vice versa within an additional 30 days, the patient will remain in the study to collect data on absolute oral bioavailability. An additional PK-curve of maximum 3 samples may be drawn.

Plasma concentrations of fluconazole will be measured in all available samples by means of a validated Liquid Chromatography with tandem mass spectrometry (LC-MS-MS) method.

A pharmacokinetic model will be fitted to the data from all individuals simultaneously. Data will be analysed using non-linear mixed effects modelling (NONMEM).After selection of the final model, a simulation study is performed using this model to assess exposure following various dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

* Subject is treated with fluconazole for prophylaxis or treatment of an invasive fungal infection;
* Subject is 2 - 18 years of age on the day of the first fluconazole dosing
* Subject is managed with a central venous catheter or arterial line from which blood can be obtained.

Exclusion Criteria:

* Subject is managed by means of an extracorporeal clearance technique;
* Subject has previously participated in this study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged 2-18 years treated with fluconazole for the prophylaxis or management of an invasive fungal infection are eligble for inclusion. In total, 30 patients will be included. Patients are treated as per local protocol. Only patients managed with a CVC or arterial line from which blood can be obtained are included to ensure the non-interventional nature of the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Target attainment of fluconazole in pediatric patients | At steady state: at day 2 after start of fluconazole therapy
  Percentage of pediatric patients reaching the predetermined pharmacokinetic/pharmacodynamic (PK/PD) target (an area-under-the-concentration-time-curve (AUC) above 400 mg*h/L)

CONTACTS AND LOCATIONS:
Overall Officials: Roger JM Brüggemann, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen
  - Prinses Máxima Centrum voor Kinderoncologie, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided